CLINICAL TRIAL: NCT00090506
Title: Yoga, Health, and Meditation
Brief Title: Yoga for Treating People at Risk for Diabetes or With Both HIV and Depression
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Center for Complementary and Integrative Health (NCCIH) (NIH)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: R21AT001942-01 (NIH)
Record Dates: First submitted 2004-08-26; First posted 2004-08-27 (Estimated); Last update posted 2008-01-25 (Estimated); Status verified 2008-01

CONDITIONS: HIV Infections; Diabetes; Depression
Keywords: Yoga; Meditation
MeSH Terms: conditions — HIV Infections; Diabetes Mellitus; Depression | interventions — Yoga

INTERVENTIONS:
Behavioral: Yoga

SUMMARY:
The purpose of this study is to plan and develop an international collaboration for research on the health effects of yoga. This study will also determine the effects of yoga on people who are at an increased risk for developing diabetes and people with both HIV and depression.

DETAILED DESCRIPTION:
In recent years, western health practitioners have become increasingly aware of the potential health benefits of yoga. This study will comprise two substudies that will evaluate the effects of yoga in two distinct populations.

Participants in the first study will be people who are at risk for developing diabetes; participants in the second study will be people with both HIV and depression. All participants will practice yoga 3 to 6 days per week for 3 months. Blood collection will be done and weight and blood pressure measurements will be taken in study 1 participants; questionnaires will be used to measure depression and stress in study 2 participants. All study participants will be assessed at entry and at 3 and 6 months.

ELIGIBILITY:
Inclusion Criteria for Study 1 Participants:

* Meet certain laboratory requirements

Inclusion Criteria for Study 2 Participants:

* HIV infected
* Able to walk at least 50% of the time

Inclusion Criteria for All Participants:

* Written informed consent of parent/guardian, if applicable

Exclusion Criteria for Study 2 Participants:

* Require antiretroviral therapy

Ages: 14 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 50
Dates: Start 2004-07; Primary Completion 2007-03 (Actual); Study Completion 2007-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Frederick M. Hecht, MD, Principal Investigator — UCSF Positive Health Program
Locations (1):
- Swami Vivekananda Yoga Anusandhana Samsthana (SVAYSA), Bangalore, India

REFERENCES:
- [Derived] McDermott KA, Rao MR, Nagarathna R, Murphy EJ, Burke A, Nagendra RH, Hecht FM. A yoga intervention for type 2 diabetes risk reduction: a pilot randomized controlled trial. BMC Complement Altern Med. 2014 Jul 1;14:212. doi: 10.1186/1472-6882-14-212. PMID 24980650